CLINICAL TRIAL: NCT03207386
Title: Preventing Sexual Violence Through a Comprehensive, Peer-led Initiative: A Process and Outcome Evaluation
Brief Title: Preventing Sexual Violence Through a Comprehensive, Peer-led Initiative
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of New Hampshire (Other)
Collaborators: Centers for Disease Control and Prevention (U.S. Federal Agency)
Responsible Party: Principal Investigator, Katie Edwards, Assistant Professor of Psychology, University of New Hampshire
Allocation: Not Applicable | Model: Sequential | Masking: None | Purpose: Prevention
Other Study IDs: UNH-03-6594&6603-01
Record Dates: First submitted 2017-06-29; First posted 2017-07-02 (Actual); Results first posted 2021-11-03 (Actual); Last update posted 2021-11-12 (Actual); Status verified 2021-11

CONDITIONS: Sexual Violence
Keywords: Sexual Violence; Prevention; Mixed-Methods; Outcome Evaluation; Process Evaluation; Adolescence

STUDY DESIGN:
Intervention Model Description: Multiple baseline survey design across three years including two baseline surveys prior to prevention programming and rollout of doses of programming across two years.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Youth VIP (Experimental): Youth VIP is a youth-led set of prevention strategies. Youth and their adult mentors are trained in evidence based sexual assault primary prevention strategies at a three day youth summit. The summit is followed by participation in working groups in which youth and their adult mentors will adapt best practices for sexual assault prevention to the Rapid City community and diffuse these strategies through both their own social networks and more formally in work in Rapid City middle and high schools.
  Interventions: Behavioral: Youth VIP

INTERVENTIONS:
Behavioral: Youth VIP — Youth VIP involves youth in partnerships with adults to adapt evidence based sexual violence prevention strategies for the local community environment. Youth VIP includes a three day intensive youth summit for prevention training and ongoing youth-adult prevention working groups.

SUMMARY:
The purpose of this multiple baseline study is to evaluate the effectiveness of a comprehensive youth-led sexual violence (SV) prevention program, Youth Voices in Prevention (Youth VIP). The prevention program builds on youth-adult partnerships among middle and high school students in Rapid City, South Dakota. Consenting students will take part in a youth summit where they will be trained as popular opinion leaders to spread SV prevention messages among middle and high school youth and parents. Following the summit, youth will work in small groups focused on different aspects of evidence-based prevention strategies including bystander intervention, social marketing messaging, parent education, norms change, and social emotional learning. Multiple research methods will be used to examine implementation process and cost. In addition, consenting students will take six surveys across three years including several surveys before programming begins, and several to document Youth VIP outcomes after prevention programming takes place. Survey data from a demographically similar community will be used to assess changes over time among youth in Rapid City, SD. All phases of the project will be implemented with collaboration from a Research Programming Advisory Board of community members and professionals from Rapid City, SD.

DETAILED DESCRIPTION:
Sexual violence (SV) impacts adolescents at rates higher than most other age demographics. Although it is a critical public health issue for youth, there are few prevention initiatives that lead to reductions in SV. There is increasing recognition that SV prevention efforts may be most effective if youth are central to the development and implementation of such efforts. Problematically, there are no rigorously evaluated youth-led SV prevention efforts, and researchers also know little about the process by which youth create prevention initiatives. Teen UP (TU) is a youth-led initiative in Rapid City, SD that focuses on addressing a variety of public health issues, including awareness about SV. This "homegrown" initiative is well integrated in the community and is the ideal platform on which additional multi-level, evidence-based SV prevention strategies can be added. Researchers and SV prevention specialists at the University of New Hampshire, in partnership with Rape Prevention Education-funded agencies in South Dakota (SD) (i.e., Network Against Family Violence and Sexual Assault [The Network] and Working Against Violence Inc. [WAVI]), will work together along with a number of community stakeholders (e.g., educators, peers, elders) and expert consultants to enhance TU to include additional SV prevention strategies, a project titled Youth Voices in Prevention (Youth VIP). Although the plan for the programming enhancement will be refined based on feedback from the Research and Programming Advisory Board (RPAB) and data collected during the refinement and planning phase of the project, the current plan is to convene a youth summit where high school youth will be trained as popular opinion leaders to diffuse SV prevention messages in addition to youth joining a formal working group specific to a SV prevention strategy that also aligns with youth's career aspirations. A mixed method approach will be used to measure implementation processes, fidelity, and costs over time, and to assess the impact of Youth VIP on rates of sexual violence perpetration among middle and high school students, as well as the secondary outcomes of sexual violence victimization, dating violence and bullying victimization and perpetration, depression, and suicidality. Collaboration with the community of students, parents, and professionals in Rapid City will be promoted by establishing a Research Programming Advisory Board (RPAB) that will meet monthly during the project.

All students in grades 7 through 10 in the fall of 2017 will be invited to participate in two baseline and four follow-up surveys that will be given in school. Surveys will take place in fall and spring of each of three school years, and the cohort enrolled in fall of 2017 will be followed over time. Recruitment of students and parents is being done in close collaboration with the Rapid City Area School District. The investigators anticipate enrolling 2,000 students.

Qualitative data includes Photovoice interviews (a technique where students take pictures of their community and describe how those pictures relate to violence in their community), interviews of students who attended programming, and interviews with key adult stakeholders. We will identify common themes in this data using content analysis, then code the interviews for these themes. We will present both the frequency that these themes emerged and key exemplary quotes. We will use a variety of methods to analyze the quantitative data. First, we will examine change in outcomes over time as a function of exposure to programming. Second, using social network analysis, we will examine change in outcomes as a function of the programming exposure of one's close friends. Third, we will use pooled cross-sectional analyses to compare students in the same grade levels over time as the program is implemented (e.g., compare this year's eight graders to last years' eighth graders). Fourth, we will use multilevel modeling to examine trajectories and changes in the cohorts (e.g., compare growth in this year's eight graders to last years' eighth graders) who are nested within schools. We will examine outcomes in these ways for primary outcome (sexual violence perpetration and victimization), intermediary outcomes (e.g., social norms), and secondary outcomes (e.g., suicidal thoughts).

ELIGIBILITY:
Inclusion Criteria:

* Must be able to complete online survey independently
* Must be a student in the Rapid City community.

Exclusion Criteria:

* None

Ages: 12 Years to 90 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 2647 (Actual)
Dates: Start 2017-02-27 (Actual); Primary Completion 2020-07-01 (Actual); Study Completion 2020-07-01 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- University of New Hampshire, Durham, New Hampshire, United States

IPD SHARING:
Plan to Share IPD: Yes

REFERENCES:
- [Background] Kann L, Kinchen S, Shanklin SL, Flint KH, Kawkins J, Harris WA, Lowry R, Olsen EO, McManus T, Chyen D, Whittle L, Taylor E, Demissie Z, Brener N, Thornton J, Moore J, Zaza S; Centers for Disease Control and Prevention (CDC). Youth risk behavior surveillance--United States, 2013. MMWR Suppl. 2014 Jun 13;63(4):1-168. PMID 24918634
- [Background] Cook-Craig PG, Coker AL, Clear ER, Garcia LS, Bush HM, Brancato CJ, Williams CM, Fisher BS. Challenge and opportunity in evaluating a diffusion-based active bystanding prevention program: Green Dot in high schools. Violence Against Women. 2014 Oct;20(10):1179-202. doi: 10.1177/1077801214551288. Epub 2014 Sep 24. PMID 25255794
- [Background] American Association of University Women. (2001) Hostile Hallways: Bullying, Teasing, and Sexual Harassment in School, American Journal of Health Education, 32:5, 307-309, DOI: 10.1080/19325037.2001.10603488
- [Derived] Edwards KM, Banyard VL, Waterman EA, Mitchell KJ, Jones LM, Kollar LMM, Hopfauf S, Simon B. Evaluating the Impact of a Youth-Led Sexual Violence Prevention Program: Youth Leadership Retreat Outcomes. Prev Sci. 2022 Nov;23(8):1379-1393. doi: 10.1007/s11121-022-01343-x. Epub 2022 Mar 18. PMID 35303249

RESULTS

PARTICIPANT FLOW:
Groups:
- Youth VIP: Youth VIP is a youth-led set of prevention strategies. Youth and their adult mentors are trained in evidence based sexual assault primary prevention strategies at a three day youth summit. The summit is followed by participation in working groups in which youth and their adult mentors will adapt best practices for sexual assault prevention to the Rapid City community and diffuse these strategies through both their own social networks and more formally in work in Rapid City middle and high schools.
  Youth VIP: Youth VIP involves youth in partnerships with adults to adapt evidence based sexual violence prevention strategies for the local community environment. Youth VIP includes a three day intensive youth summit for prevention training and ongoing youth-adult prevention working groups.
  Participants could be in both the large camp condition and/or the small camp condition, thus numbers do not consistently add up to 2647 across the results reports for the study.
Period: Overall Study
Arm/Group | Youth VIP
Started | 2647
Completed | 1487
Not Completed | 1160

BASELINE CHARACTERISTICS:
Arm/Group | Youth VIP
Number analyzed (Participants) | 2647
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 2647
  Between 18 and 65 years | 0
  >=65 years | 0
Sex/Gender, Customized [Count of Participants; unit: Participants]
  Sex at Birth: Female | 1355
  Sex at Birth: Male | 1269
  Sex at Birth: Unknown | 23
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 334
  Not Hispanic or Latino | 2239
  Unknown or Not Reported | 74
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 410
  Asian | 38
  Native Hawaiian or Other Pacific Islander | 30
  Black or African American | 58
  White | 1823
  More than one race | 259
  Unknown or Not Reported | 29
Region of Enrollment [Number; unit: participants]
  United States | 2647

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants Reporting Any Form of Sexual Violence Perpetration
Description: We used several measures to assess for a wide range of interpersonal violence victimization perpetration experiences during the past six months, all with response options 1 = yes or 0 = no. Outcome counts indicate number of participants who reported yes to any form of sexual violence perpetration. We used mirror items to assess for both victimization and perpetration experiences. Three items assessing sexual assault were drawn from Cook-Craig et al.'s (2014) measure that assessed for sexual coercion, physically-forced sex, and incapacitated sex. Five items from the YRBS were used to assess physically forced sexual contact, sexual dating violence, physical dating violence, bullying on school property, and electronic bullying (Centers for Disease Control and Prevention, 2014). We used three items from the American Association of University Women (2001) to assess homophobic teasing, sexual harassment, and sexual rumors. Lastly, two items assessed homophobic bullying and racial bullying.
Time Frame: 6 months
Population: Participants could be in both the large camp condition and/or the small camp condition, thus numbers do not consistently add up to 2647 across the results reports for the study.
Measure: Count of Participants; unit: Participants
Groups:
- Attended Large Camp: Participants attended a large prevention camp.
- Did Not Attend Large Camp: Participants did not attend a large prevention camp.
- Attended Small Camp: Participants attended a small prevention camp.
- Did Not Attend Small Camp: Participants did not attend a small prevention camp.
Arm/Group | Attended Large Camp | Did Not Attend Large Camp | Attended Small Camp | Did Not Attend Small Camp
Number analyzed (Participants) | 104 | 2434 | 81 | 2457
Participants | 5 | 54 | 2 | 57

2. Secondary Outcome: Number of Participants Reporting Any Form of Sexual Violence Victimization
Description: We used several measures to assess for a wide range of interpersonal violence victimization perpetration experiences during the past six months, all with response options 1 = yes or 0 = no. Outcome counts indicate number of participants who reported yes to any form of sexual violence victimization. We used mirror items to assess for both victimization and perpetration experiences. Three items assessing sexual assault were drawn from Cook-Craig et al.'s (2014) measure that assessed for sexual coercion, physically-forced sex, and incapacitated sex. Five items from the YRBS were used to assess physically forced sexual contact, sexual dating violence, physical dating violence, bullying on school property, and electronic bullying (Centers for Disease Control and Prevention, 2014). We used three items from the American Association of University Women (2001) to assess homophobic teasing, sexual harassment, and sexual rumors. Lastly, two items assessed homophobic bullying and racial bullying.
Time Frame: 6 months
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Attended Large Camp | Did Not Attend Large Camp | Attended Small Camp | Did Not Attend Small Camp
Number analyzed (Participants) | 104 | 2434 | 81 | 2457
Participants | 13 | 97 | 6 | 104

ADVERSE EVENTS:
Time Frame: Adverse events were collected over thirty months.
Arm/Group | Youth VIP
All-Cause Mortality (participants affected / at risk) | 0/2647
Serious Adverse Events (participants affected / at risk) | 0/2647
Other Adverse Events (participants affected / at risk) | 0/2647

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (3):
  • Study Protocol (2021-08-19): https://cdn.clinicaltrials.gov/large-docs/86/NCT03207386/Prot_001.pdf
  • Statistical Analysis Plan (2021-08-19): https://cdn.clinicaltrials.gov/large-docs/86/NCT03207386/SAP_002.pdf
  • Informed Consent Form (2019-07-29): https://cdn.clinicaltrials.gov/large-docs/86/NCT03207386/ICF_000.pdf